CLINICAL TRIAL: NCT01144507
Title: Prediction by Ultrasound of the Risk of Hepatic Cirrhosis in Cystic Fibrosis (PUSH)
Brief Title: Prediction by Ultrasound of the Risk of Hepatic Cirrhosis in Cystic Fibrosis
Acronym: PUSH
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CFLD PUSH; U01DK062456 (NIH)
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis; Pancreatic Insufficiency
Keywords: Cystic Fibrosis; Pancreatic insufficiency
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During this study, blood and urine specimens will be obtained, de-identified and shipped to and stored at the NIDDK repositories for use in future CFLD ancillary studies. This "biobanking" is a critical aspect of this longitudinal study to facilitate the creation of a resource of DNA and other specimens from a meaningful number of patients with CFLD. In addition, obtaining and storing DNA or EBV-transformed leukocytes (from which DNA can be extracted) will allow future studies to investigate genetic causes and influences (modifier genes) in CFLD.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group A: Approximately 60 subjects with a heterogeneous echo pattern of the liver on abdominal ultrasound (HTG US).
  Interventions: Procedure: Abdominal Ultrasound; Other: Sample collection procedures
- Group B: Approximately 680 subjects with a normal echo pattern on abdominal ultrasound (NL US). Of these subjects, approximately 110 will be matched 1:1 with Group A participants and followed for the duration of the study. The remaining unmatched subjects will not be followed beyond their initial visit.
  Interventions: Procedure: Abdominal Ultrasound; Other: Sample collection procedures
- Group C: An estimated 30 subjects with cirrhosis pattern on abdominal ultrasound. These subjects will be followed in the study.
  Interventions: Procedure: Abdominal Ultrasound; Other: Sample collection procedures
- Group D: An estimated 30 subjects with diffusely homogeneous echogenic pattern at screening ultrasound will be followed in the study.
  Interventions: Procedure: Abdominal Ultrasound; Other: Sample collection procedures

INTERVENTIONS:
Procedure: Abdominal Ultrasound — To establish eligibility and/or markers regarding echo pattern types.
  Other Names: Doppler Ultrasound
Other: Sample collection procedures — Samples of urine, serum, plasma, and blood for DNA from children and blood for DNA from parents will be requested from participating subjects
  Other Names: Doppler Ultrasound

SUMMARY:
The specific aims for this study are:

1. To determine if sonographic findings predict the risk of progression of liver disease to cirrhosis by comparing cystic fibrosis subjects with heterogeneous echogenicity pattern on ultrasound to those with normal echogenicity pattern on ultrasound
2. To develop a database and biorepository of serum, plasma, urine and DNA to aid the investigations in ascertaining the mechanisms, consequences, genetic risk factors and biomarkers for the development of cirrhosis
3. To determine if there are differences in health related quality of life, pulmonary or nutritional status in children with cystic fibrosis who have a heterogeneous echo pattern on ultrasound compared to those who have a normal echo pattern on ultrasound
4. To determine if Doppler velocity measurements of hepatic and splenic vessels predict an increased risk for the development of cirrhosis.
5. To determine if cirrhosis on ultrasound progresses to portal hypertension during the study period
6. To determine if homogeneous liver progresses to either cirrhosis or heterogeneous liver.
7. To determine the frequency of complications of portal hypertension during follow up in those identified with cirrhosis by year 6 of the study

DETAILED DESCRIPTION:
For subjects in longitudinal follow up, this study will:

1. Collect detailed clinical and demographic information about each subject at enrollment and during follow up,
2. Obtain and store imaging data from the subject at entry and during follow up,
3. Obtain and store serum, plasma and urine samples from the subject at entry (after matching) and during follow up,
4. Obtain and store DNA from the subject,
5. Obtain and store DNA from the biological parents,
6. Obtain and store quality of life data from the subject and parents at enrollment and during follow up

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 through 12 years of age at time of enrollment diagnosed with Cystic Fibrosis and pancreatic insufficiency
* Enrolled in the CFF registry study or Toronto CF Registry
* CF defined as sweat chloride of >60 mEq/L on one occasion (using the value in the CF registry) or two disease-causing mutations of CFTR with evidence of end organ involvement.
* Pancreatic insufficient defined as one of the following:

  * CFTR Mutation associated with pancreatic insufficiency
  * Fecal elastase <100 mcg/gm (at any time)
  * 72 hour fecal fat with coefficient of fat absorption <85% (at any time)

Exclusion Criteria:

* Known cirrhosis
* Presence of Burkholderia cepacia
* Short bowel syndrome defined as not on full enteral feeds by 3 months of age
* Presence of other serious disease precluding participation in this study (This would include patients with known other causes of chronic liver disease)
* If in the opinion of the Investigator the study is not in the best interest of the patient
* Inability to comply with the longitudinal follow-up described below
* Failure of a family to sign the informed consent document or the HIPAA medical record release form

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of males and females 3 through 12 years of age with Cystic Fibrosis and pancreatic insufficiency who are enrolled in the CFF or Toronto CF registry studies. All racial and ethnic groups will be included.
Sampling Method: Non-Probability Sample
Enrollment: 774 (Actual)
Dates: Start 2010-01-12 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Development of cirrhosis, as defined by imaging criteria | Nine years
  The primary objective of this prospective longitudinal study is to determine the utility of abdominal ultrasound (US) at enrollment to predict the development of cirrhosis in subjects with cystic fibrosis (CF) within a nine year period.

SECONDARY OUTCOMES:
Effects on associated pulmonary and nutritional issues | 9years
  * Health related quality of life
  * Growth (length, weight and BMI Z-score, anthropometrics)
  * AST,ALT,GGTP
  * FEV1, FVC
  * Sputum Culture (Pseudomonas, Burkholderia cepacia)
  * Use of IV antibiotics
  * Hospitalization for treatment of pulmonary exacerbation
  * CBC (WBC, Hbg, ANC, platelet count)
  * Fat soluble vitamin levels (Vitamin E, 25 hydroxy vitamin D, Vitamin A)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Narkewicz, MD, Study Chair — Children's Hospital Colorado; Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Averell Sherker, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (11):
- United States (10):
  - Children's Hospital of Colorado, Aurora, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - University of Minneapolis Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Siegel MJ, Freeman AJ, Ye W, Palermo JJ, Molleston JP, Paranjape SM, Stoll J, Leung DH, Masand P, Karmazyn B, Harned R, Ling SC, Navarro OM, Karnsakul W, Alazraki A, Schwarzenberg SJ, Seidel FG, Towbin A, Alonso EM, Nicholas JL, Murray KF, Otto RK, Sherker AH, Magee JC, Narkewicz MR; CFLD Network. Heterogeneous Liver on Research Ultrasound Identifies Children with Cystic Fibrosis at High Risk of Advanced Liver Disease: Interim Results of a Prospective Observational Case-Controlled Study. J Pediatr. 2020 Apr;219:62-69.e4. doi: 10.1016/j.jpeds.2019.12.033. Epub 2020 Feb 12. PMID 32061406
- [Derived] Siegel MJ, Leung DH, Molleston JP, Ye W, Paranjape SM, Freeman AJ, Palermo JJ, Stoll J, Masand P, Karmazyn B, Harned R, Ling SC, Navarro OM, Karnsakul W, Alazraki A, Schwarzenberg SJ, Towbin AJ, Alonso EM, Nicholas JL, Green N, Otto RK, Magee JC, Narkewicz MR. Heterogeneous liver on research ultrasound identifies children with cystic fibrosis at high risk of advanced liver disease. J Cyst Fibros. 2023 Jul;22(4):745-755. doi: 10.1016/j.jcf.2023.03.019. Epub 2023 Apr 7. PMID 37032248
- [Derived] Leung DH, Ye W, Molleston JP, Weymann A, Ling S, Paranjape SM, Romero R, Schwarzenberg SJ, Palermo J, Alonso EM, Murray KF, Marshall BC, Sherker AH, Siegel MJ, Krishnamurthy R, Harned R, Karmazyn B, Magee JC, Narkewicz MR; Cystic Fibrosis Liver Disease Network (CFLD NET). Baseline Ultrasound and Clinical Correlates in Children with Cystic Fibrosis. J Pediatr. 2015 Oct;167(4):862-868.e2. doi: 10.1016/j.jpeds.2015.06.062. Epub 2015 Aug 5. PMID 26254836
- See also: PUSH is a study in the ChiLDREN Network — http://www.childrennetwork.org/